CLINICAL TRIAL: NCT01725971
Title: The Use of Forced Oscillation Technique in the Analysis of Respiratory System in Never-smoking Patients With Silicosis:Pathophysiological Study and Evaluation of Diagnostic Accuracy
Brief Title: Oscillation Mechanics of the Respiratory System in Never-smoking Patients With Silicosis
Status: Completed | Type: Observational
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Paula Morisco de Sá, researcher, Rio de Janeiro State University
Other Study IDs: Silicose2012; Silicose2012 (Other: UERJ)
Record Dates: First submitted 2012-10-30; First posted 2012-11-14 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Silicosis
Keywords: Silicosis; forced oscillations; respiratory mechanics
MeSH Terms: conditions — Silicosis

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Control group: Group of nonsmokers individuals without respiratory disease.
- normal exam: subjects with silicosis , but with normal spirometric data
- mild obstruction: subjects with silicosis with mild obstruction in spirometric data
- moderate to severe obstruction: subjects with silicosis with moderate to severe obstruction in spirometric data

SUMMARY:
Silicosis is a chronic and incurable occupational disease that can progress independent of the end of exposure. Recent works suggest that the Forced Oscillation Technique (FOT) may help to improve our understanding of the changes in lung mechanics, as well as in the detection of these changes.

Objectives: Analyze the effects of airway obstruction in silicosis on the respiratory impedance and evaluated the diagnostic use of the FOT in these patients. For this, the investigators used spirometry to classify airway obstruction, which resulted in four categories: control, patients with normal exam, mild obstruction, and moderate-to-severe obstruction. Resistive data were interpreted using the zero-intercept resistance (R0), the resistance at 4 Hz (Rrs4) and the mean resistance (Rm). The investigators also analyzed the mean reactance (Xm) and the dynamic compliance (Crs,dyn). The total mechanical load was evaluated using the absolute value of the respiratory impedance (Z4Hz). The diagnostic potential was evaluated by investigating the area under the receiver operating characteristic curve (AUC).

ELIGIBILITY:
Inclusion Criteria:

* • Volunteers with silicosis for Patients Group;

  * Volunteers without any respiratory disease for the control group.

Exclusion Criteria:

* Smokers

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The control group will consist of healthy subjects, nonsmokers, who had no episode of respiratory infection thirty days before the examinations.
  The group with diagnosis of silicosis was established based on a history of substantial exposure to silica dusts and compatible radiological features, together with exclusion of other competing diagnoses.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2010-07; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
spirometric | 1 day
  Spirometry was used to classify airway obstruction, which resulted in four categories: control (n=21), patients with normal exam (n=12), mild obstruction (n=22), and moderate-to-severe obstruction (n=12).
Forced Oscillation technique | 1 day
  In the analysis of the forced oscillation technique was used the following data: Resistive data were interpreted using the zero-intercept resistance (R0), the resistance at 4 Hz (Rrs4) and the mean resistance (Rm). The researchers also analyzed the mean reactance (Xm) and the dynamic compliance (Crs,dyn). The total mechanical load was evaluated using the absolute value of the respiratory impedance (Z4Hz).

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratório de Instrumentação Biomédica, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Sa PM, Lopes AJ, Jansen JM, Melo PL. Oscillation mechanics of the respiratory system in never-smoking patients with silicosis: pathophysiological study and evaluation of diagnostic accuracy. Clinics (Sao Paulo). 2013 May;68(5):644-51. doi: 10.6061/clinics/2013(05)11. PMID 23778400